CLINICAL TRIAL: NCT03888339
Title: Influence of Different Abutment Shape on Peri-implant Marginal Bone Loss: A Randomized Clinical Trial.
Brief Title: Influence of Abutment Shape on Peri-implant Marginal Bone Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Peñarrocha Oltra, Assistanat Postdoctoral Lecturer (Profesor Ayudante Doctor), University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H1524219380739
Record Dates: First submitted 2018-12-11; First posted 2019-03-25 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Dental Implant; Bone Resorption
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group - Commercially available high abutments (Active Comparator): Commercially available 2.5mm high abutments
  Interventions: Procedure: Commercially available high abutments placement
- Test group - Modified shape abutments (Experimental): Modified shape 2.5mm high abutments (imitating the shape of 0.5mm short abutments)
  Interventions: Procedure: Modified shape abutments

INTERVENTIONS:
Procedure: Commercially available high abutments placement — Patients will be randomly selected for the commercially available high abutments option. Two or three implants will be placed following the drilling protocol suggested by the manufacturer. Implants will be placed 0.5mm subcrestal. Once the implants have been placed, periapical radiographs and clinical pictures will be taken. Implants will be uncovered 10 weeks after being placed. After performing the incision and elevation a minimal flap, conventional high transmucosal abutments will be screwed using the torque recommended by the manufacturer. Once the abutments have been screwed, periapical radiographs and clinical pictures will be taken. The abutments will not be unscrewed thereafter throughout the study.
  Arms: Control group - Commercially available high abutments
Procedure: Modified shape abutments — Patients will be randomly selected for the modified shape abutments option. Two or three implants will be placed following the drilling protocol suggested by the manufacturer. Implants will be placed 0.5mm subcrestal. Once the implants have been placed, periapical radiographs and clinical pictures will be taken. Implants will be uncovered 10 weeks after being placed. After performing the incision and elevation a minimal flap, modified high transmucosal abutments will be screwed using the torque recommended by the manufacturer. Once the abutments have been screwed, periapical radiographs and clinical pictures will be taken. The abutments will not be unscrewed thereafter throughout the study.
  Arms: Test group - Modified shape abutments

SUMMARY:
A study designed as a randomized controlled trial of parallel group design will be conducted at the Dental clinic of the University of Valencia to evaluate the influence of 2.5 mm high abutments with different shapes (commercially available high abutments vs high abutments with modified shape to imitate short abutments) on peri-implant bone loss around bone level implants with platform switching in partially edentulous patients that require a fixed rehabilitation supported by two implants in the posterior mandible or maxilla and in fixed rehabilitation supported by one implant in the anterior mandible or maxilla.

DETAILED DESCRIPTION:
A study designed as a randomized controlled trial of parallel group design will be conducted at the Dental clinic of the University of Valencia to evaluate the influence of 2.5 mm high abutments with different shapes (commercially available high abutments vs high abutments with modified shape to imitate short abutments) on peri-implant bone loss around bone level implants with platform switching in partially edentulous patients that require a fixed rehabilitation supported by two implants in the posterior mandible or maxilla and in fixed rehabilitation supported by one implant in the anterior mandible or maxilla (from premolar to premolar).

ELIGIBILITY:
Inclusion Criteria:

* Any subject requiring two implants in the posterior mandible or maxilla, being at least 18 years old and able to sign an informed consent. Final patient inclusion will be made after flap elevation during the implant placement surgery to be able to confirm the presence of a vertical thickness ≥ 3mm of keratinized soft tissues.
* Bone volumes should allow the placement of implants at least 8 mm long (i.e, 10 mm bone height to the inferior alveolar nerve) and 4.2 mm wide (7 mm wide bone crest) without bone regeneration procedures.
* Patients will be grouped into: 1) non smokers; 2) light smokers (≤ 10 cigarettes/day); 3) heavy smokers (≥ 11 cigarettes/day)

Exclusion Criteria:

* Patients unable to commit to follow-up.
* General contraindications to implant surgery.
* Immuno-suppressed/immune-compromised patients.
* Patients irradiated in the head and/or neck.
* Uncontrolled diabetes.
* Pregnancy or lactation.
* Untreated periodontal disease.
* Poor oral hygiene and motivation.
* Addiction to alcohol or drugs.
* Psychiatric problems and/or unrealistic expectations.
* Patients with an acute infection (abscess) or suppuration in the site intended for implant placement.
* Patients treated or under treatment with intravenous amino-bisphosphonates.
* Patients referred only for implant placement if the follow-up cannot be done at the treatment center.
* Patients participating in other studies, if the present protocol could not be fully adhered to.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Peri-implant bone level changes | 12 months after implant loading
  Assessed on digital periapical radiographs taken with the paralleling technique at delivery of crowns (implant loading) and 12 months afterwards.

SECONDARY OUTCOMES:
Implant survival rate | 12 months after implant loading
  % of implants in function
Probing pocket depth | 12 months after implant loading
  Measured in millimeters with a millimetered periodontal probe
Bleeding on probing | 12 months after implant loading
  Positive or negative bleeding after having probed with a millimetered periodontal probe
Peri-implant soft tissue recession | 12 months after implant loading
  Measured in millimeters with a millimetered periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Odontológica de la Universitat de Valencia, Fundación Lluis Alcanyis, Valencia, Spain